CLINICAL TRIAL: NCT03108196
Title: A Multicenter Randomized Controlled Study to Compare the Safety and Efficacy of Detaenial Sigmoid Neobladder and Hautmann Ileal Neobladder in Patients with Bladder Cancer
Brief Title: Comparison of Safety and Efficacy of Detaenial Sigmoid Neobladder and Ileal Neobladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Sun Yat-sen University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Fourth Affiliated Hospital of Guangxi Medical University (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Abai Xu, Chief, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2016PY030
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer; Urinary Diversion
Keywords: bladder cancer， neobladder, detaenial sigmoid, ileal
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Superiority verification based on the ileal neobladder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sigmoid (Experimental): Use 15 cm detaenial sigmoid colon to reconstructed a "U" shape neobladder after radical cystectomy.
  Interventions: Procedure: sigmoid
- ileal (Experimental): Use 70 cm distal ileal segment to reconstructed a "spherical" shape neobladder after radical cystectomy.
  Interventions: Procedure: ileal

INTERVENTIONS:
Procedure: sigmoid — The serosal layer with smooth muscle was detached from a 15 cm sigmoid segment submucosal layer and removed continuously. Only the mucosal and submucosal layers were preserved. Approximately 2 cm of the taeniae and serosal layer were preserved to strengthen the urethra-neobladder anastomosis at the central portion of the isolated sigmoid and at the two ends for the ureter-neobladder anastomosis. The ureters were subsequently implanted in antirefluxing fashion in a submucosal tunnel. The ureter-neobladder anastomoses were protected with a 6Fr Single J® stent. The two ends of the sigmoid were closed with the embedded seromuscular layer. The neobladder was anastomosed to the urethra after that.
  Arms: sigmoid
Procedure: ileal — The isolated 70 cm terminal ileum segment is arranged in either an M or W shape and is opened along the antimesenteric border except for a 5 cm section where the incision is curved to make a U-shaped ﬂap. The four limbs of the M or W are then sutured to one another with a running absorbable suture. A small full-thickness segment of bowel is excised for the urethral anastomosis. Once the ileal neobladder is situated and the urethral sutures are tied, the ureters are implanted from inside the neobladder through a small incision in the ileum. The remaining portion of the anterior wall is then closed with a running absorbable suture. Ureteroileal anastomosis were performed with a freely refluxing, open end-to-side method at each end of the W.
  Arms: ileal

SUMMARY:
Bladder cancer is a common malignant tumor of the urinary system, radical resection plus urinary diversion is the first choice of treatment for muscle invasive bladder cancer. Urinary diversion of surgical options related to patient' survival and quality of life.

In 1988, Hautmann firstly reported an orthotopic urinary diversion method: Hautmann neobladder. As the urine can be controlled from the original urethra, the patient's quality of life has been greatly improved, so the new bladder surgery gradually accepted and welcomed by urologists and patients. However, in order to achieve low-pressure and large-volume storage capacity of the urine reservoir, the 40-70cm long interception of terminal ileum need to be detubularized. Only after split, folded, re-stitched and a series of treatment, the intestinal can be used. Such complicated procedures make so many urologists give it up. In addition, the interception of the long ileum may lead to reduced absorption of vitamin B12 which caused anemia, metabolic acidosis, intestinal dysfunction. Not only that, as time goes by, this kind of neobladder will be unlimited expansion and resulting in a serious increase in residual urine volume, hydronephrosis, or even the occurrence of neobladder spontaneous rupture.

In 2000, professor Chunxiao Liu invented "detaenial sigmoid neobladder", this surgical method overset the traditional intestinal detubularization approach, which detached the serosal layer with smooth muscle from the bowel without split it. This kind of neobladder is easier to construct and have less impact on intestinal function. So far, it has been implemented for more than 600 cases in Zhujiang hospital, the age of patients range from 9 months (bladder rhabdomyosarcoma) to 84 years old.

So far as now, no multicenter prospective clinical study on orthotopic urinary diversion has been performed worldwide, neither the head-to-head studies on detaenial sigmoid neobladder and ileal neobladder.

Our project is going to perform a multicenter randomized controlled trial for these two neobladder methods and look forward to assess the safety and efficacy of these two procedures which provide an objective basis for the patients undergoing orthotopic urinary diversion in the future.

DETAILED DESCRIPTION:
Surgical technique for Hautmann ileal neobladder: A 70-cm portion of terminal ileum is selected and incised on the antimesenteric border. The ileum is arranged into an M or W configuration with the four limbs sutured to one another. After a buttonhole of ileum is removed on an antimesenteric portion of the ileum, the urethral anastomosis is performed. The ureteral anastomoses are performed using a Le Duc technique or direct implantation, are stented, and the reservoir is then closed in a side-to-side manner. As an alternative, the two ends of the W may be left slightly longer as a short chimney on either side for implantation of the ureters.

Surgical technique for detaenial sigmoid neobladder: After radical cystectomy, the sigmoid was brought out from a midline incision in the lower abdomen and a 15 to 25 cm segment was isolated. Intestinal continuity was restored using a circular stapler. Omental and free taeniae, and the serosal layer were incised deeply as far as the submucosal layer until the plane between smooth muscle and the submucosal layer could be identified clearly by scalpel dissection. The serosal layer with smooth muscle was then detached from the submucosal layer and removed continuously without difficulty. During this time, the operator could insert the finger in the sigmoid lumen and lift the sigmoid wall up for accurate dissection. Only the mucosal and submucosal layers were preserved. Approximately 2 to 3 cm of the taeniae and serosal layer were preserved to strengthen the urethra-neobladder anastomosis at the central portion of the isolated sigmoid and at the two ends for the ureter-neobladder anastomosis. The detaenial sigmoid was irrigated repeatedly by dilute iodine solution to eliminate impurities. Its capacity for enlargement and leak tightness were assessed at the end by filling with 300 to 400 ml iodine solution. Residual taeniae were identified and incised during this filling phase. The ureters were subsequently implanted in antirefluxing fashion in a submucosal tunnel with 4-zero poly glactin at the two ends of sigmoid. The ureter-neobladder anastomoses were protected with a 6Fr Single J® stent. Each stent was passed through the sigmoid wall and exteriorized. The two ends of the sigmoid were closed by 2-zero polyglactin with the embedded seromuscular layer. The central portion of the sigmoid was incised and a 22Fr 3-way catheter was inserted in neobladder. The neobladder was anastomosed to the urethra with 2-zero polyglactin.

Followup: Each patient was evaluated at 3-month intervals for 1 year, at 6-month intervals for 2 to 5 years. Renal ultrasound, biochemical examination and urine culture were done every 3 to 6 months. Pelvic computerized tomography and retro-cystogram were performed 6 months postoperatively and annually thereafter. Urodynamic investigation and cystoscopic examination were done annually.

Postoperative complications were classified as early (90 days or less) and late (greater than 90 days). Early and late complications were subdivided into those related and not related to the neobladder. Complication grade was classified according to the Clavien-Dindo system. Major complications were defined as grade III or higher. Daytime and nighttime continence levels were recorded postoperatively at patient interview. Continence was defined as complete if the patient was dry without a pad, satisfactory if no more than 1 pad was required and poor if the patient used more than 1 pad during the day or night.

End points: The primary end point was change in renal function from baseline to 3 years. Secondary end points included changes in renal function from baseline to 6, 12 and 24 months, reduction in eGFR 10 ml/minute/1.73 m2 or greater, early (less than 90 days) and late (90 days to 3 years) complications, urinary tract infection that was symptomatic or was treated, any surgical re-intervention or urinary diversion related surgical re-intervention defined as an open or endoscopic procedure under anesthesia, cancer recurrence and overall survival. Renal function was assessed using the CKD-EPI equation. Complications were analyzed and graded by a blinded adjudicator using the modified Clavien complication grading system.

ELIGIBILITY:
Inclusion Criteria:

1. Bladder carcinoma in situ, include CIS and T1G3 tumor, muscle invasive bladder cancer（T2/T3N0-1M0）
2. Recurrent bladder cancer
3. Other conditions that have been approved by a urologist for indications for new bladder surgery
4. Had been received intravesical chemotherapy, intra-arterial infusion chemotherapy or systemic chemotherapy in the past.
5. Voluntarily signed the informed consent -

Exclusion Criteria:

1. Preoperative serum creatinine more than 2.26mg/dl（Or 200μmol/L）
2. Cancer invaded urethral (confirmed by the pathology)
3. Non - bladder cancer patients underwent neobladder
4. A history of other malignant tumors within five years
5. Ileum / sigmoid chronic inflammation, like ulcerative colitis or intestinal tuberculosis, and so on.
6. Other conditions that have been approved by a urologist for not suitable for new bladder surgery

   -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Post void residual volume of neobladder | the 36th month
  Residual urine volume after spontaneous urination with urinary diversion in the 36th month

SECONDARY OUTCOMES:
Time cost | 24 hour
  Time consuming of neobladder construction
EBL | 24 hour
  Estimated blood loss
Short term complications | 90 day postoperative
  Complications which happened during 90 day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Abai Xu, doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All released data will be available for other researchers.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Witjes JA, Comperat E, Cowan NC, De Santis M, Gakis G, Lebret T, Ribal MJ, Van der Heijden AG, Sherif A; European Association of Urology. EAU guidelines on muscle-invasive and metastatic bladder cancer: summary of the 2013 guidelines. Eur Urol. 2014 Apr;65(4):778-92. doi: 10.1016/j.eururo.2013.11.046. Epub 2013 Dec 12. PMID 24373477
- [Background] Hautmann RE, Egghart G, Frohneberg D, Miller K. The ileal neobladder. J Urol. 1988 Jan;139(1):39-42. doi: 10.1016/s0022-5347(17)42283-x. PMID 3336101
- [Background] Zerhau P, Husar M. [Mucus production consequences in cystoplasties and continent urinary diversions in children--long term experiences]. Rozhl Chir. 2006 Mar;85(3):148-50. Czech. PMID 16689148
- [Background] Haupt G, Pannek J, Knopf HJ, Schulze H, Senge T. Rupture of ileal neobladder due to urethral obstruction by mucous plug. J Urol. 1990 Sep;144(3):740-1. doi: 10.1016/s0022-5347(17)39571-x. PMID 2388342
- [Background] Xu K, Liu CX, Zheng SB, Li HL, Xu YW, Xu AB, Chen BS, Shen HY. Orthotopic detaenial sigmoid neobladder after radical cystectomy: technical considerations, complications and functional outcomes. J Urol. 2013 Sep;190(3):928-34. doi: 10.1016/j.juro.2013.03.072. Epub 2013 Mar 26. PMID 23538237
- [Background] Xu A, Li B, Li H, Zheng S, Du W, Xu Y, Zou Y, Luo Q, Liu C. Comparison of seromuscular tunnel and split-cuff nipple antireflux ureteroenteral anastomosis techniques in orthotopic taenia myectomy sigmoid neobladder: a prospective, randomized study. Urology. 2013 Mar;81(3):669-74. doi: 10.1016/j.urology.2012.11.018. Epub 2013 Jan 3. PMID 23290142
- [Background] Skinner EC, Fairey AS, Groshen S, Daneshmand S, Cai J, Miranda G, Skinner DG. Randomized Trial of Studer Pouch versus T-Pouch Orthotopic Ileal Neobladder in Patients with Bladder Cancer. J Urol. 2015 Aug;194(2):433-9. doi: 10.1016/j.juro.2015.03.101. Epub 2015 Mar 28. PMID 25823791
- [Background] Bacchetti P, Leung JM. Sample size calculations in clinical research. Anesthesiology. 2002 Oct;97(4):1028-9; author reply 1029-32. doi: 10.1097/00000542-200210000-00050. No abstract available. PMID 12357184
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Miyake H, Furukawa J, Sakai I, Muramaki M, Yamashita M, Inoue TA, Fujisawa M. Orthotopic sigmoid vs. ileal neobladders in Japanese patients: a comparative assessment of complications, functional outcomes, and quality of life. Urol Oncol. 2013 Oct;31(7):1155-60. doi: 10.1016/j.urolonc.2011.11.015. Epub 2011 Dec 6. PMID 22153716
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912